CLINICAL TRIAL: NCT06927102
Title: A Comprehensive Analysis of Follow-up Outcomes, Continuity and Updated Survivorship in Breast Cancer
Brief Title: From Exclusion to Inclusion: Analysing Follow-up Discontinuity in Breast Cancer
Acronym: FOCUS-BC
Status: Recruiting | Type: Observational
Sponsor: Basavatarakam Indo American Cancer Hospital & Research Institute (Other)
Responsible Party: Principal Investigator, Nisha Hariharan, Consultant, Breast Oncosurgeon, Basavatarakam Indo American Cancer Hospital & Research Institute
Other Study IDs: IEC/2024/295
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Carcinoma
Keywords: Breast cancer; Follow up; survivorship
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- New, non-metastatic, breast cancer patients between 2017-2018: All women with newly diagnosed non-metastatic breast cancer, presenting to Basavatarakam Indo American Cancer Hospital & Research Institute, Hyderabad, India, between 2017 - 2018 will be included in the study. The analysis will focus on the women who have been lost-to-follow-up.

SUMMARY:
The goal of this observational study is to determine the proportion of patients who are lost-to-follow-up at five years, identify factors associated with loss of follow-up , and explore patient-reported barriers to follow-up in a public sector cancer care setting.

The main question it aims to answer is : Do proactive outreach programs help in improving follow-up rates among breast cancer patients who are categorized as "lost-to-follow-up." This study will be conducted in a real-world cohort of women with non-metastatic breast cancer treated at a tertiary care centre, between 2017-2018.

DETAILED DESCRIPTION:
This is a prospective cohort study involving women diagnosed with non-metastatic breast cancer in the years 2017-2018, who received treatment at our institute. Baseline data collection will include essential demographic information, clinical data including tumor characteristics, stage at presentation and luminal subtype and treatment information including surgical intervention, chemotherapy, radiotherapy, hormonal therapy, and targeted therapy.

The study will be conducted in three phases.

1. Phase I: Quantitative Follow-Up Analysis Follow-up data will be retrieved from hospital records and electronic medical records (EMR) up to December 2024. Follow-up visits will be documented annually through to the end of 2024.
2. Phase II: Assessment of Lost to Follow-Up (LTFU) Cases For patients identified as LTFU (definitions provided below), additional variables will be extracted, including geographic distance from the hospital, mode of employment, marital status, and payment method (government scheme, insurance, or self-pay). Proactive outreach efforts will be undertaken via phone calls, messages, or emails using contact information available in hospital records. Informed consent will be obtained in cases where contact has been successfully established - verbally for phone calls and in writing for electronic communication. Patients (or their families) will be queried about current health status, recent diagnostic evaluations, recurrence of disease, or mortality (if applicable). These responses will be documented as valid follow-up entries.
3. Phase III: Qualitative Analysis of LTFU Reasons During outreach, participants will also be asked to identify reasons for missing follow-up visits. These will be categorized under the following domains: Logistical barriers (e.g., travel, time constraints), financial constraints, availability of alternative/local healthcare facilities, physician recommendations, lack of awareness regarding the importance of follow-up. In addition, participants will be asked about their willingness to maintain hospital contact in the future and their preferred mode of communication (e.g., phone, SMS, email, video call).

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly diagnosed with non-metastatic breast cancer between 2017-2018
2. Patients categorized as "lost-to-follow-up", as defined above
3. Patients willing to participate upon re-engagement

Exclusion Criteria:

1. Patients with incomplete medical records
2. Patients who have taken part of the treatment at another hospital/centre
3. Patients who have relocated permanently out of the study region

Withdrawal Criteria:

1. Patient withdraws consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective cohort study involving women diagnosed with non-metastatic breast cancer in the years 2017-2018, who received treatment at our institute, Basavatarakam Indo American Cancer Hospital & Research Institute, Hyderabad, India.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in follow-up data with proactive outreach | 6 months
  Follow-up data will be retrieved from hospital records and electronic medical records (EMR) up to December 2024. For patients identified as lost-to-follow-up, proactive outreach efforts will be undertaken via phone calls, messages, or emails. Patients (or their families) will be queried about recurrence of disease, and these responses will be documented as valid follow-up entries.
Updated mortality data | 6 months
  For patients identified as lost-to-follow-up, proactive outreach efforts will be undertaken via phone calls, messages, or emails. Patients (or their families) will be queried about mortality (if applicable) and these responses will be documented as valid follow-up entries.

SECONDARY OUTCOMES:
3. Evaluate the reasons for patient disengagement from follow-up care. | 6 months
  During outreach, participants will also be asked to identify reasons for missing follow-up visits. These will be documented as qualitative entries.
Assessment of willingness for future hospital contact | 6 months
  Participants will be asked about their willingness to maintain hospital contact in the future and their preferred mode of communication.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Hariharan, MS,HBNI Fellow Breast Oncology, Principal Investigator — Basavatarakam Indo American Cancer Hospital & Research Institute
Locations (1):
- Basavatarakam Indo American Cancer Hospital & Research Institute, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Undecided
Since this study involves contacting women who are lost-to-follow-up, the investigators are considering various options for sharing IPD, with appropriate consent from the participants.

REFERENCES:
- [Derived] Hariharan N, Rao TS, Rajappa SJ, Naidu CK, Rayani B, Kodandapani S, Koppula V, Gudipudi D. From exclusion to inclusion: Analysis of patterns of follow-up in breast cancer. Int J Surg Protoc. 2025 Sep 8;29(4):156-160. doi: 10.1097/SP9.0000000000000061. eCollection 2025 Dec. PMID 41334423